CLINICAL TRIAL: NCT06781970
Title: The Effects of Vitamin C Supplementation on Corneal Endothelial Damage in Hard Cataract Phacoemulsification: an Oxidative Stress Study on Aqueous Humour and Corneal Endothelial Cell Characteristics.
Brief Title: Effect of Vitamin C Supplementation in Corneal Endothelial Damage in Phacoemulsification of Patients with Hard Cataracts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Melva Louisa, Prof. dr. Melva Louisa, S.Si., M.Biomed, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-08-1198
Record Dates: First submitted 2024-12-17; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Endothelial Cell Loss, Corneal; Cataract and Intraocular Lens (IOL) Surgery
Keywords: Cataract; Corneal Endothelial Damage; Phacoemulsification; Total Antioxidant Capacity; Ascorbic Acid; Vitamin C Supplementation; malondialdehyde
MeSH Terms: conditions — Corneal Endothelial Cell Loss; Cataract; Intraocular Lymphoma | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vit C (Experimental): Patient will consume 500 mg of oral vitamin C, tid, 7 days prior to phacoemulsification to 4 weeks after phacoemulsification
  Interventions: Drug: Oral Vitamin C
- Preoperative Vit C (Experimental): Patient will consume 500 mg of oral vitamin C, tid, 7 days prior to phacoemulsification and placebo, tid, 4 weeks after phacoemulsification
  Interventions: Drug: Oral Vitamin C; Drug: Placebo
- Placebo (Placebo Comparator): Patient will consume placebo, tid, 7 days prior to phacoemulsification to 4 weeks after phacoemulsification
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Vitamin C — Patients will be given 500 mg of oral vitamin C, tid, for 7 days prior to phacoemulsification and 4 weeks after phacoemulsification
  Other Names: ascorbic acid
  Arms: Preoperative Vit C; Vit C
Drug: Placebo — Patients will be given placebo, tid, for 7 days prior to phacoemulsification and 4 weeks after phacoemulsification
  Arms: Placebo; Preoperative Vit C

SUMMARY:
The goal of this clinical trial is to analyze the protective effects of oral ascorbic acid on the corneal endothelial layer undergoing oxidative stress due to phacoemulsification in patients with hard cataracts. The main questions it aims to answer are:

1. Will oral vitamin C administration provide better protection to the corneal endothelium in hard cataract phacoemulsification by comparing preoperative and postoperative administration, preoperative only, and no administration?
2. How does oxidative stress (MDA levels) in the aqueous humour increase after oral vitamin C administration compared to no administration?
3. Will there any changes in MDA levels in the aqueous humour and blood after oral vitamin C administration compared to no administration?
4. Does MDA levels in the aqueous humour correlate with MDA levels in the blood?

Researchers will compare vitamin C to a placebo to see if vitamin C as an antioxidant works in preventing corneal endothelial damage due to phacoemulsification.

Participants will:

* Take 500 mg of oral vitamin C or placebo three times a day for seven days prior to phacoemulsification
* Undergo phacoemulsification
* Take vitamin C or placebo three times a day for 28 days after phacoemulsification
* Visit the ophthalmology clinic 1, 7, 28, and 42 days post-operative for checkups
* Keep a logbook to record the drug they take and to write symptoms of possible side effect of the drug

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 60 years or older
* Patients with immature senile cataracts in one or both eyes, with LOC (lens opacities classification) III nuclear opacity grade 4-6 and nuclear color grade 4-6 criteria
* Patients willing to undergo phacoemulsification cataract surgery and consume the study medication as allocated, as well as participate in follow-up assessments for 7 weeks
* Patients with no history of previous intraocular surgery
* Patients with no history of allergy to vitamin C
* Patients not routinely consuming other vitamins
* Patients who agree to and sign the informed consent for the study

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Endothelial cell loss | From the start of the study to six weeks after intervention
  Difference of endothelial cell density before and after phacoemulsification

SECONDARY OUTCOMES:
Serum ascorbic acid levels | From the start of the study to seven days after intervention
  Level of ascorbic acid in serum
Serum total antioxidant capacity levels | From the start of the study to seven days after intervention
  Level of total antioxidant capacity in serum
Serum malondialdehyde levels | From the start of the study to seven days after intervention
  Levels of malondialdehyde in serum
Aqueous ascorbic acid levels | Right before phacoemulsification
  Level of aqueous ascorbic acid
Aqueous total antioxidant capacity levels | Right before phacoemulsification
  Levels of total antioxidant capacity in aqueous humour
Aqueous malondialdehyde levels | Right before phacoemulsification to 3 minutes after phacoemulsification
  Levels of malondialdehyde in aqueous humour
Central corneal thickness | rom the start of the study to six weeks after intervention
  Thickness of the central part of the cornea
Grading of cells in anterior chamber | From the start of the study to six weeks after intervention
  Collection of white blood cells in the anterior chamber
Visual acuity of patients | From the start of the study to six weeks after intervention
  A measure of the ability of the eye to distinguish shapes and the details of objects at a given distance

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Pharmacology Laboratory of the University of Indonesia, Jakarta, DKI Jakarta
  - RSUD Sayang, Cianjur, West Java

IPD SHARING:
Plan to Share IPD: No
Protection of patient data and privacy